CLINICAL TRIAL: NCT00657410
Title: Randomized Study of the Treatment of Primary Immune Thrombocytopenic Purpura (ITP) in Newly Diagnosed Untreated Adult Patients. Comparison of Standard Dose Prednisone Versus High-dose Dexamethasone.
Brief Title: Prednisone or Dexamethasone in Newly Diagnosed, Previously Untreated Primary Immune Thrombocytopenic Purpura
Acronym: ITP0207
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP0207; GIMEMA-ITP-0207; Eudract 2008-000417-30; EU-20839
Record Dates: First submitted 2008-04-11; First posted 2008-04-14 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Nonneoplastic Condition
Keywords: idiopathic thrombocytopenic purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A - PDN (Experimental): PDN is administered orally at the daily dose of 1 mg/Kg for 4 consecutive weeks (from day 0 to day 28), then, therapy is tapered within 14 days. The patients considered NOT RESPONDER at day 42 or WHO HAVE LOST THE RESPONSE within the evaluation of final response (see paragraph 8.1), will be crossed to ARM B.
  Interventions: Drug: prednisone; Procedure: quality-of-life assessment
- ARM B - DXM (Experimental): DXM is administered orally at single fixed daily doses of 40 mg for 4 consecutive days, every 14 days, for 3 consecutive courses. If platelet count is £ 20x109/L or bleeding symptoms related to thrombocytopenia are present, lowdose DXM (0.035 mg/Kg/day) between courses is given. The patients (either from ARM A+B or from ARM B) considered NOT RESPONDER at day 46 or who HAVE LOST THE RESPONSE within the evaluation of final response (see paragraph 8.1), will be considered OFF TREATMENT.
  For these patients a second line therapy will be considered, according to the medical practice of the Centre (splenectomy or other).
  Interventions: Drug: dexamethasone; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: dexamethasone
  Arms: ARM B - DXM
Drug: prednisone
  Arms: ARM A - PDN
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs, such as prednisone and dexamethasone, may change the immune system and be an effective treatment for primary immune thrombocytopenic purpura. It is not yet known which drug is more effective in treating primary immune thrombocytopenic purpura.

PURPOSE: This randomized phase III trial is studying high-dose dexamethasone to see how well it works compared to standard-dose prednisone in treating patients with newly diagnosed, previously untreated primary immune thrombocytopenic purpura.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the role of therapy intensification in adult patients with newly diagnosed, previously untreated primary immune thrombocytopenic purpura with high-dose dexamethasone (HD-DXM), in terms of improvement of response at 6 months after initial response, in comparison with standard-doses of prednisone.

Secondary

* Compare rate of initial response.
* Compare quality of response.
* Compare rate of final responses and rate of persistent response.
* Compare rate of bleeding events.
* Determine rate of resumed response with HD-DXM in non-responder patients or patients who have lost response (arm I only).
* Compare time to platelet number increase until a hemostatically effective level is reached and/or disappearance of bleeding symptoms.
* Compare rate of rescue interventions.
* Compare rate of eligible patients for splenectomy.
* Compare rate of patients who underwent splenectomy.
* Compare rate of patients who develop connective tissue diseases or underlying hematological diseases (myelodysplastic syndromes, chronic lymphoproliferative diseases, others).
* Compare patient's self reported quality of life.

OUTLINE: This is a multicenter study. Patients are stratified by treating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (Standard-dose prednisone): Patients receive oral prednisone at a standard dose (1 mg/Kg) once daily on days 1-28 followed by a 14-day taper.

Patients considered non-responders at day 42 or who have lost response before evaluation of final response (day 180) are crossed to arm II.

* Arm II (High-dose dexamethasone): Patients receive oral dexamethasone at a high dose (40 mg/day) once daily on days 1-4. Treatment repeats every 14 days for 3 courses.

Quality of life is assessed at baseline, on day 42 (arm I) or 46 (arm II) (initial response evaluation day), 180 days after initial response evaluation, and at 3, 9, 12 months after randomization.

After completion of study treatment, patients are followed monthly until 1 year after randomization, every 2 months for 1 year, and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion criteria

* Signed written informed consent according to IGH/EU/GCP and national local laws
* Newly diagnosed untreated ITP adult patients
* Age > 18 < 80 years
* Platelet count <20x109/L
* Platelet count > 20 x109/L and <50x109/L plus bleeding with score > 8 (according to grading scale at paragraph 7.1)
* Baseline Quality of Life evaluation questionnaire filled in Newly diagnosed untreated ITP adult patients
* Age > 18 < 80 years
* Platelet count <20x109/L
* Platelet count > 20 x109/L and <50x109/L plus bleeding with score > 8 (according to grading scale at paragraph 7.1)
* Baseline Quality of Life evaluation questionnaire filled in

Exclusion criteria

* Active malignancy at time of study entry
* Steroids administration (PDN <1mg/Kg/day) for more than 5 days before randomization
* Concomitant treatment with anti-platelet and or anti-coagulant drugs
* Concomitant severe psychiatric disorders
* Not confirmed diagnosis of ITP for

  * *Positivity of autoimmunity markers: antinucleus (≥1:80), anti-tireoglobulin, anti-tireoperoxidase, anti-cardiolipin (≥ 40 GPL UmL), anti-b2glycoprotein (≥ 40 IgG U/mL) antibodies, Lupus Anticoagulant (KCT ratio, dRVVT ratios ≥1.5 times the upper normal limit ), direct antiglobulin test (DAT ).
  * Presence of autoimmune hemolytic anemia
  * Presence of connective tissue disease
* Women who are pregnant or breastfeeding
* Cardiovascular diseases requiring treatment
* Severe non-controlled, despite therapy, hypertension and diabetes
* Liver and kidney function impairment (creatinine, ALT, AST >2 times upper normal limit)
* HCVAb, HIVAb, HBsAg, HBcAb seropositive status
* Chronic liver disease
* Documented viral illness by the positivity of IgM, or vaccination both occurred one month before diagnosis
* Intake of drugs not previously taken within one week before diagnosis
* Bleeding score 15 due to ICH or to GI bleeding (according to grading scale at paragraph 7.1, Tab. 3)
* Active gastric ulcer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Final response (complete, partial, and minimal response) rate from evaluation of initial response | At day +180 from evaluation of initial response

SECONDARY OUTCOMES:
Initial response rate | At day 42 (arm I), at day 46 (arm II)
Quality of response per arm | At initial evaluation and at final evaluation
Final response rate | At day 180 from the statement of initial response
Rate of bleeding events | At 3 years from study entry
Resumed response rate in non-responder patients (at day 42) or patients who have lost response before day 180 from the first evaluation (arm I only) | At day 42 or before day 180 from the first evaluation
Time to platelet number increase until a hemostatically effective level is reached and/or disappearance of bleeding symptoms | At 3 years from study entry
Rate of persistent response | At 12 months from the statement of initial response
Association of type of initial response with final and persistent response (in patients with final and persistent response) | At 3 years from study entry
Rate of rescue interventions | After day 180 from evaluation of initial response
Rate of splenectomy eligible patients | At 12 months from enrollment
Rate of patients who have undergone splenectomy during follow-up | At 3 years from study entry
Rate of patients who develop connective tissue diseases or underlying hematological diseases (myelodysplastic syndromes, chronic lymphoproliferative diseases, others) during follow-up | At 3 years from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gabriella Mazzucconi, MD, Principal Investigator — Gruppo Italiano Malattie EMatologiche dell'Adulto
Locations (42):
- Italy (42):
  - U.O. di Ematologia - Azienda Ospedaliera - Pia Fondazione di Culto e di Religione Card. G.Panico, Tricase, (le)
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda ospedaliera Nuovo Ospedale "Torrette", Ancona
  - USL 8 - Ospedale S.Donato, Arezzo
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - UO Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - University of Bologna Medical School, Bologna
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Struttura Complessa di Oncologia Medica - Azienda Ospedaliera - Ospedale di Circolo di Busto Arsizio, Busto Arsizio
  - Marche U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Marche
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Ospedale Maggiore - Div.Medicina Crema, Crema
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Ospedale Santa Maria Goretti, Latina
  - ASL Le1 P.O. Vito Fazzi - U.O. di Ematologia, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Azienda Ospedaliera San Paolo - Unità di Ematologia e Trombosi, Milan
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Med. Int. ed Oncologia Medica IRCCS Policlinico S. Matteo, Pavia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Pordenone Unità operativa Medicina II Az. Osp. S. M. degli Angeli, Pordenone
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - UOC Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Struttura Complessa II Medicina - Ematologia - Centro di Riferimento Ematologico - Ospedale Maggiore, Trieste
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Policlinico G. B. Rossi - Borgo Roma, Verona
  - Ospedale San Bortolo, Vicenza

REFERENCES:
- [Derived] Mazzucconi MG, Rodeghiero F, Avvisati G, De Stefano V, Gugliotta L, Ruggeri M, Vianelli N, Fazi P, Paoloni F, Sargentini V, Baldacci E, Ferretti A, Martino B, Vincelli ID, Carli G, Fortuna S, Di Ianni M, Ranalli P, Palandri F, Polverelli N, Lugli E, Rivolti E, Patriarca A, Rago A, D'Adda M, Gentile M, Siragusa S, Sibilla S, Carella AM, Rossi E, Battistini R, Zaja F, Bocchia M, Di Renzo N, Musto P, Crugnola M, Giuffrida AC, Krampera M, Tafuri A, Santoro C. Prednisone vs high-dose dexamethasone in newly diagnosed adult primary immune thrombocytopenia: a randomized trial. Blood Adv. 2024 Mar 26;8(6):1529-1540. doi: 10.1182/bloodadvances.2023010975. PMID 38231017